CLINICAL TRIAL: NCT05412654
Title: Testing the Potential Effect of a Potassium-rich Water Intervention on Blood Pressure in Mild to Moderately Hypertensive Adults: a Double-blind Randomised Controlled Trial
Brief Title: Potassium Supplementation to Reduce Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Collaborators: Suntory Beverage & Food Limited (Unknown)
Responsible Party: Principal Investigator, Shelly Coe, Senior Lecturer in Nutrition, Oxford Brookes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 221579
Record Dates: First submitted 2022-05-31; First posted 2022-06-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Prehypertension
Keywords: Potassium; Blood pressure; Systolic; Randomised
MeSH Terms: conditions — Prehypertension; Systolic Murmurs

STUDY DESIGN:
Intervention Model Description: Double blinded randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High potassium water (Experimental): All participants will be provided with bottled water for the duration of the 4 week intervention to consume 1L/day. The intervention group will receive high potassium water. Participants will be instructed to consume 1 bottle (500 mL) within 2 hours after waking up and 1 bottle (500 mL) within 2 hours before going to bed (total 1L/day). Participants will continue with the same diet and exercise patterns in their daily life similar to before participating in the study, for the whole length of the intervention.
  Interventions: Dietary Supplement: High potassium water
- Low potassium control water (Placebo Comparator): All participants will be provided with bottled water for the duration of the 4 week intervention to consume 1L/day. The control group will receive regular bottled mineral water. Participants will be instructed to consume 1 bottle (500 mL) within 2 hours after waking up and 1 bottle (500 mL) within 2 hours before going to bed (total 1L/day). Participants will continue with the same diet and exercise patterns in their daily life similar to before participating in the study, for the whole length of the intervention.
  Interventions: Dietary Supplement: Control low potassium water

INTERVENTIONS:
Dietary Supplement: High potassium water — High potassium water Potassium 6.2 mg/100ml
  Arms: High potassium water
Dietary Supplement: Control low potassium water — Control water Potassium 0.2 mg/100ml
  Arms: Low potassium control water

SUMMARY:
The aim of this study is to conduct a definitive trial to assess the efficacy of consuming 1L/day of water rich in potassium to reduce blood pressure in mild to moderately hypertensive adults. The objective is to assess the potential effect of the intervention on reducing systolic blood pressure. This study will comprise of a 4 week, double-blind, parallel randomised controlled trial. Participants will be adults with systolic blood pressure measurements of 130mmHg or greater. The intervention comprises advice to consume bottled water rich in potassium. The comparator will be regular bottled mineral water.This study will recruit 40 people with elevated systolic blood pressure (≥130mmHg) who are not regularly taking antihypertensive medication.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Between 20 to 64 years old
* English speaking
* Adults who are not receiving antihypertensive pharmacological treatment
* Recent (within 6 months) and latest systolic blood pressure measurement ≥130mmHg and/or diastolic ≥85 mmHg
* Have access to internet and equipment for video calling
* Able to post samples and equipment to OxBCNH
* Physically able to take own body measurements and blood pressure

Exclusion Criteria:

* Participation in another research study
* Unable to read and understand the instructions provided in English
* Unable to comply with experimental procedures or not follow testing safety guidelines
* People with cardiovascular conditions: heart attack or stroke within the last 3 months, heart failure of grade II New York Heart Association and more severe, or prolonged QT syndrome, angina, arrhythmia or atrial fibrillation.
* Uncontrolled type 2 diabetes (HbA1c> 9%)
* Type 2 diabetes controlled using exogenous insulin
* Previous or current diagnosis of diabetes complications such as nephropathy, retinopathy and neuropathy.
* People with type 1 diabetes
* Currently on any medication that may lead to hyperkalemia or fluid retention
* Currently being assessed for diagnosis of hypertension (not receiving treatment for high blood pressure)
* Already on clinician/HCP supervised diet or restricted diet
* They are planning on going away from home (holiday or other) during the 4 week intervention period and will not be able to take water during this time.
* Currently prescribed antihypertensive medications, or have been in the last 6 weeks
* Chronic kidney disease stage 1 (G1A2 or G1A3), 2 (G2A2 or G2A3), 3a, 3b, 4 or 5 based on UKKA (we will ask whether participants have been diagnosed with kidney disease by a clinician based on this criteria)
* They are planning to go on a diet or begin taking supplements containing potassium during the intervention
* Pregnant women (including women suspected of being pregnant) and breast-feeding woman.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Seated home measured systolic blood pressure mm/Hg | Blood pressure will be taken at three time points through out the 4 weeks.
  Blood pressure will me monitored by the participant at home, after detailed instruction are provided by trained researchers over Zoom. Measurements will be taken in duplicate, in the morning and again in the evening (4 times a day total) and the average values will be taken.

SECONDARY OUTCOMES:
Seated home measured diastolic blood pressure | Blood pressure will be taken at three time points through out the 4 weeks
  Blood pressure will me monitored by the participant at home, after detailed instruction are provided by trained researchers over Zoom. Measurements will be taken in duplicate, in the morning and again in the evening (4 times a day total) and the average values will be taken.
Qualitative semi-structured, part open ended survey of acceptability of trial and reported barriers | This survey will be administered on the final visit at week 4 of the trial.
  This survey will be designed by the researchers understand the participant experience of the intervention, in order to optimise any future study expansion. This will include things that worked well and those that did not work as well, during the trial (consumption of the water, convenience, appropriateness of outcome measures, burden on daily activities and lifestyle, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No